CLINICAL TRIAL: NCT00648908
Title: Phase 3 Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR in Subjects With Multiple Sclerosis Who Participated in the MS-F203 Trial
Brief Title: Open-Label Extension Study to Evaluate the Safety, Tolerability and Activity of Oral Fampridine-SR Tablets in Multiple Sclerosis Patients Who Participated in the MS-F203 Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-F203EXT
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MS; walking; leg strength; demyelination
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fampridine-SR — Tablets, 10 mg, BID
  Other Names: 4-aminopyridine

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and activity of Fampridine-SR when administered for up to 36 additional months, or until it becomes commercially available whichever comes first, in subjects who previously participated in Acorda Therapeutics Protocol MS-F203.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a disorder of the body's immune system that affects the central nervous system (CNS). Normally, nerve fibers carry electrical impulses through the spinal cord, providing communication between the brain and the arms and legs. In people with MS, the fatty sheath that surrounds and insulates the nerve fibers (called "myelin") deteriorates, causing nerve impulses to be slowed or stopped. As a result, patients with MS may experience periods of muscle weakness and other symptoms such as numbness, loss of vision, loss of coordination, paralysis, spasticity, mental and physical fatigue and a decrease in the ability to think and/or remember. These periods of illness may come (exacerbations) and go (remissions). Fampridine-SR is an experimental drug that has been reported to possibly improve muscle strength and walking ability for some people with MS. This study will evaluate the effects and possible risks of taking Fampridine-SR in MS patients over a long period of time.

ELIGIBILITY:
Inclusion Criteria:

* subject must have been previously enrolled in Acorda Therapeutics MS-F203 study for multiple sclerosis and received either Fampridine-SR or placebo
* subject is a man or woman with clinical definite multiple sclerosis as defined by McDonald (McDonald WI, et al. Recommended Diagnostic Criteria for Multiple Sclerosis; Guidelines from the International Panel on the Diagnosis of Multiple Sclerosis; Annals of Neurology. 2001; 50: 121-127)
* subject must be at least 18 years of age. Any subject who is now over the age of 70 must be in good overall health in the judgment of the Investigator
* subject must be of adequate cognitive function, as judged by the Investigator, to understand and sign the IRB/REB-approved informed consent form prior to the performance of any study-specific procedures and is willing to comply with the required scheduling and assessments of the protocol
* subjects who are women of childbearing potential, regardless of sexual activity, must have a negative urine pregnancy test at the Screening Visit.

Exclusion Criteria:

* women who are either pregnant or breastfeeding, and women of childbearing potential (defined as not surgically sterile or at least two years post menopausal) who are engaged in active heterosexual relations and, are not using one of the following birth control methods: tubal ligation, implantable contraception device, oral, patch, injectable or transdermal contraceptive, barrier method or sexual activity restricted to vasectomized partner.
* subject discontinued prematurely from the MS-F203 study
* subject has a history of seizures or has evidence of past, or possible, epileptiform activity on an EEG
* subject has either a clinically significant abnormal ECG or laboratory value(s) at the Screening visit, as judged by the Investigator that would preclude entry into the study. ECG and laboratory results from Visit 6 or repeat results from Visit 7 of the MS-F203 study may be used as the baseline for the current study
* subject has angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality, as judged by the Investigator
* subject has a known allergy to pyridine-containing substances or any of the inactive ingredients of the Fampridine-SR tablet (hydroxypropyl methylcellulose, microcrystalline cellulose, colloidal silicon dioxide, magnesium stearate, opadry white (tablet film coating))
* subject has received an investigational drug, except for Fampridine-SR or matching placebo under protocol MS-F203, within 30 days of the Screening Visit. Subject is scheduled to enroll in an investigational drug trial at any time during this study.
* subject has a history of drug or alcohol abuse within the past year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2006-06; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Faust, Study Director — Acorda Therapeutics
Locations (32):
- United States (27):
  - Barrow Neurology Clinic, St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC, Keck School of Medicine Health Care Consultation Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - Shepherd Center, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University MS Center, Indianapolis, Indiana
  - Maryland Center for MS, Baltimore, Maryland
  - Wayne State University, Department of Neurology, Detroit, Michigan
  - The Schapiro Center for MS, Golden Valley, Minnesota
  - Washington University School of Medicine, Div. of Rehab/Neurology, St Louis, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - Gimbel MS Center at Holy Name Hospital, Teaneck, New Jersey
  - Maimonides MS Care Center, Brooklyn, New York
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - CMC - Neuroscience & Spine Institute, Division of Neurology, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University MS Center, Columbus, Ohio
  - Oregon Health & Science University, MS Center of Oregon, UHS-42, Portland, Oregon
  - Thomas Jefferson University Physicians, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - University of Texas-Houston, Houston, Texas
  - Neurological Research Center, Inc., Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - MS Center at Evergreen, Kirkland, Washington
- Canada (5):
  - Foothills Medical Center, Calgary, Alberta
  - University of British Columbia, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - River Valley Health c/o Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - QEII Health Sciences Centre, Nova Scotia Rehabilitation Centre Site, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario

REFERENCES:
- See also: (Click here for more information about Fampridine-SR clinical trials) — http://www.acorda.com/clinical.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Fampridine-SR: Tablets, 10mg twice daily
Period: Overall Study
Arm/Group | Fampridine-SR
Started | 269
Completed | 154
Not Completed | 115

BASELINE CHARACTERISTICS:
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 256
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 52.1 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 251
  More than one race | 3
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment Emergent Adverse Events (TEAE).
Description: All adverse events reported were treatment emergent. Therefore, events that had a date of onset, or worsening, on or after the start of the open-label drug and up to 14 days after the last dose (for non-serious events) or up to 30 days after the last dose (for SAEs) were summarized. Any abnormal clinically significant changes in physical examination, medical history, clinical laboratory testing, 12-lead ECG, and standard EEG testing were captured as adverse events.
Time Frame: up to 5 years
Population: Safety Population. No imputation for missing data
Measure: Number; unit: Participants
Arm/Group | Fampridine-SR 10mg (Twice a Day)
Number analyzed (Participants) | 269
Participants
  Patients with Any TEAE | 264
  Patients with Any Serious AE | 94
  Patients with Any Possibly/Probably Related AE | 77
  Patients Withdrawn due to AE | 37
  Patients who Died | 4
  Maximum Severity /Patients with Any Mild TEAE | 16
  Maximum Severity /Patients with Any Moderate TEAE | 137
  Maximum Severity /Patients with Any Severe TEAE | 111

2. Secondary Outcome: Timed 25 Foot Walk (T25FW)
Time Frame: Week 2, 14, 26, continuing every 26 weeks until the Final Visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Fampridine-SR 10mg (Twice a Day)
Number analyzed (Participants) | 267
feet/second
  (N=265) >0-8 Weeks | 2.35 (0.96)
  (N=242) >8-16 Weeks | 2.27 (0.95)
  (N=249) >16-42 Weeks | 2.28 (1.02)
  (N=222) >42-68 Weeks | 2.23 (1.10)
  (N=204) >68-94 Weeks | 2.18 (1.05)
  (N=190) >94-120 Weeks | 2.15 (1.00)
  (N=177) >120-146 Weeks | 2.14 (1.03)
  (N=156) >146-172 Weeks | 2.14 (0.99)
  (N=143) >172-198 Weeks | 2.14 (1.06)
  (N=137) >198-224 Weeks | 2.15 (1.05)
  (N=58) >224-250 Weeks | 1.98 (1.09)
  (N=7) >250-276 Weeks | 1.56 (0.97)

3. Secondary Outcome: Subject Global Impression (SGI)
Description: Patients asked to complete a Subject Impression questionnaire rating his/her impression of the effects of study drug during the preceding week, specifically in regards to signs and symptoms associated with Multiple Sclerosis (MS).
  For the SGI, the potential responses to the effects of the investigational drug during the preceding week were 1=terrible, 2=unhappy, 3=mostly dissatisfied, 4=neutral/ mixed, 5=mostly satisfied, 6=pleased, and 7=delighted.
Time Frame: visit 1 and every clinic visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 268
units on a scale
  (N=268) >0-8 Weeks | 4.85 (1.10)
  (N=247) >8-16 Weeks | 4.79 (1.12)
  (N=247) >16-42 Weeks | 4.86 (1.19)
  (N=230) >42-68 Weeks | 4.80 (1.28)
  (N=214) >68-94 Weeks | 4.95 (1.20)
  (N=203) >94-120 Weeks | 5.03 (1.18)
  (N=191) >120-146 Weeks | 5.14 (1.14)
  (N=182) >146-172 Weeks | 5.09 (1.05)
  (N=168) >172-198 Weeks | 5.13 (1.11)
  (N=159) >198-224 Weeks | 5.16 (1.07)
  (N=77) >224-250 Weeks | 5.20 (1.01)
  (N=13) >250-276 Weeks | 5.46 (1.13)

4. Secondary Outcome: Clinician Global Impression of Change (CGIC)
Description: Investigator's overall impression of the patients neurological status and general state of health related to his/her participation in the study; specifically signs and symptoms associated with MS.
  The potential responses were 1=very much improved, 2=much improved, 3=somewhat improved, 4=no change, 5=somewhat worse, 6=much worse, and 7=very much worse.
Time Frame: visit 1 and every clinic visit
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 267
units on a scale
  (N=267) >0-8 Weeks | 3.38 (0.88)
  (N=248) >8-16 Weeks | 3.56 (0.98)
  (N=256) >16-42 Weeks | 3.55 (0.87)
  (N=233) >42-68 Weeks | 3.63 (0.99)
  (N=215) >68-94 Weeks | 3.66 (0.98)
  (N=203) >94-120 Weeks | 3.59 (0.99)
  (N=194) >120-146 Weeks | 3.69 (1.01)
  (N=179) >146-172 Weeks | 3.85 (1.02)
  (N=167) >172-198 Weeks | 3.75 (1.08)
  (N=160) >198-224 Weeks | 3.93 (1.13)
  (N=76) >224-250 Weeks | 3.97 (1.34)
  (N=13) >250-276 Weeks | 3.39 (1.12)

5. Secondary Outcome: Expanded Disability Status Scale (EDSS)
Description: Each patient, based on their baseline neurological exam, are scored according to the EDSS
  The EDSS was used to grade patient disability on a scale from 0.0 (normal neurological exam) to 10.0 (death) at the Screening Visit, Visit 6, and Final Visit or Early Termination Visit if applicable.
Time Frame: Screening visit, visit 6 and every 24 months thereafter
Population: ITT Population. No imputation for missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fampridine-SR
Number analyzed (Participants) | 268
units on a scale
  (N=268) Baseline | 5.78 (1.07)
  (N=192) >94-120 Weeks | 5.95 (1.13)
  (N= 148) >198-224 Weeks | 6.16 (0.94)

ADVERSE EVENTS:
Arm/Group | Fampridine-SR
Serious Adverse Events (participants affected / at risk) | 94/269
Other Adverse Events (participants affected / at risk) | 264/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fampridine-SR (N=269)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Affective Disorder (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1)
Aphagia (Gastrointestinal disorders) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bacterial Pyelonephritis (Infections and infestations) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candida Sepsis (Infections and infestations) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 5 (6)
Cellulitis Staphylococcal (Infections and infestations) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Cervical Cord Compression (Nervous system disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Clostridial Infection (Infections and infestations) | 1 (1)
Clostridium Colitis (Infections and infestations) | 3 (3)
Completed Suicide (Psychiatric disorders) | 1 (1)
Complex Partial Seizures (Nervous system disorders) | 1 (1)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Device Failure (Injury, poisoning and procedural complications) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 3 (3)
Hyperparathyroidism Primary (Endocrine disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 (2)
Major Depression (Psychiatric disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Medical Observation (Investigations) | 1 (1)
Menorrhagia (Renal and urinary disorders) | 1 (1)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 13 (19)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasticity (Nervous system disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous System Disorder (Nervous system disorders) | 1 (1)
Neurogenic Bladder (Renal and urinary disorders) | 1 (2)
Nodal Rhythm (Cardiac disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Open Wound (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Parvovirus Infection (Infections and infestations) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Abscess (Infections and infestations) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Splenic Rupture (Injury, poisoning and procedural complications) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tracheal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (8)
Urinary Tract Infection Staphylococcal (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 3 (3)
Varicose Vein Ruptured (Vascular disorders) | 1/1 (1)
Volvulus of Bowel (Gastrointestinal disorders) | 1 (1)
Vulvar Dysplasia (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fampridine-SR (N=269)
Adverse Drug Reaction (General disorders) | 22 (37)
Anxiety (Psychiatric disorders) | 16 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 66 (93)
Asthenia (General disorders) | 41 (50)
Back Pain (Musculoskeletal and connective tissue disorders) | 45 (56)
Balance Disorder (Nervous system disorders) | 18 (20)
Blood Cholesterol Increased (Investigations) | 14 (17)
Cellulitis (Infections and infestations) | 15 (20)
Constipation (Gastrointestinal disorders) | 27 (30)
Contusion (Injury, poisoning and procedural complications) | 31 (46)
Cystitis (Infections and infestations) | 28 (62)
Depression (Psychiatric disorders) | 38 (50)
Diarrhoea (Gastrointestinal disorders) | 28 (38)
Dizziness (Nervous system disorders) | 28 (35)
Fall (Injury, poisoning and procedural complications) | 107 (291)
Fatigue (General disorders) | 44 (56)
Headache (Nervous system disorders) | 28 (39)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 18 (18)
Hypoaesthesia (Nervous system disorders) | 26 (35)
Influenza (Infections and infestations) | 19 (26)
Insomnia (Psychiatric disorders) | 40 (45)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 20 (23)
Multiple Sclerosis (Nervous system disorders) | 21 (24)
Multiple Sclerosis Relapse (Nervous system disorders) | 87 (160)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 34 (45)
Muscle Spasticity (Nervous system disorders) | 42 (49)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 35 (44)
Nasopharyngitis (Infections and infestations) | 37 (56)
Nausea (Gastrointestinal disorders) | 40 (60)
Oedema Peripheral (General disorders) | 53 (66)
Pain (General disorders) | 21 (24)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 53 (71)
Paraesthesia (Nervous system disorders) | 25 (36)
Pollakiuria (Renal and urinary disorders) | 15 (15)
Pyrexia (General disorders) | 17 (22)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 19 (25)
Sinusitis (Infections and infestations) | 26 (45)
Skin Laceration (Injury, poisoning and procedural complications) | 17 (19)
Tremor (Nervous system disorders) | 14 (15)
Upper Respiratory Tract Infection (Infections and infestations) | 47 (70)
Urinary Incontinence (Renal and urinary disorders) | 15 (15)
Urinary Tract Infection (Infections and infestations) | 112 (319)
Vomiting (Gastrointestinal disorders) | 18 (24)
White Blood Cell Count Increased (Investigations) | 14 (17)
White Blood Cells Urine Positive (Investigations) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.